CLINICAL TRIAL: NCT02808390
Title: A Phase 2, Randomized, Placebo-controlled, Multicenter Study to Investigate the Efficacy and Safety of GED-0507-34-Levo (GED0507) for Treatment of Subjects With Active Ulcerative Colitis
Brief Title: Efficacy and Safety Study of GED-0507-34-Levo for Treatment of UC
Acronym: SEGMENT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: PPM Services S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GED0507-UC-001
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 80 mg BID (Experimental): GED-0507-34-Levo 80 mg BID for 8 Weeks
  Interventions: Drug: GED-0507-34-Levo 80 mg
- 160 mg BID (Experimental): GED-0507-34-Levo 160 mg BID for 8 Weeks
  Interventions: Drug: GED-0507-34-Levo 160 mg
- Placebo (Experimental): Placebo BID for 8 Weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GED-0507-34-Levo 80 mg — GED-0507-34-Levo 80 mg BID for 8 Weeks
  Arms: 80 mg BID
Drug: GED-0507-34-Levo 160 mg — GED-0507-34-Levo 160 mg BID for 8 Weeks
  Arms: 160 mg BID
Drug: Placebo — Placebo BID for 8 Weeks
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of 2 doses of GED-0507-34-Levo in subjects with active, mild-to-moderate UC.

DETAILED DESCRIPTION:
This is a Phase 2, Proof of Concept, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of 2 doses of GED-0507-34-Levo in subjects with active, mild-to-moderate Ulcerative Colitis.

The study will consist of 3 phases:

* Screening Phase - up to 4 weeks
* Double-blind Placebo-controlled Phase - Weeks 0 to 8
* Follow-up Phase - Week 9

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over at the time of signing the informed consent.
* Diagnosis of UC with a duration of at least 3 months prior to the Screening Visit.
* MMS ≥ 4 to ≤ 8 (range: 0 - 9) prior to randomization in the study
* Subjects are required to have a colonoscopy if one has not been performed within 12 months prior to the Screening Visit.
* Subjects who have relapsed on maintenance therapy with doses of 5-ASA ≤ 2.4 g/day

Exclusion Criteria:

* Diagnosis of Crohn's disease, indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis, or diverticular disease-associated colitis.
* UC restricted to the distal 15 cm or less (eg, ulcerative proctitis).
* Subjects who have had surgery as a treatment for UC or who, in the opinion of the Investigator, are likely to require surgery for UC during the study.
* Clinical signs suggestive of fulminant colitis or toxic megacolon.
* Evidence of pathogenic enteric infection.
* History of colorectal cancer or colorectal dysplasia.
* Prior use of any TNF inhibitor (or any biologic agent).
* Prior use of mycophenolic acid, tacrolimus, sirolimus, cyclosporine, or thalidomide.
* Use of budesonide-MMx within the last 8 weeks.
* Use of oral and/or IV corticosteroids within 2 weeks of the Screening Visit.
* Use of immunosuppressants (azathioprine [AZA], 6-mercaptopurine [6-MP] or methotrexate [MTX]) within 8 weeks of the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (11):
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Center for Advanced Gastroenterology, PLLC, Maitland, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - IMIC, Inc, Palmetto Bay, Florida
  - BRCR Medical Center, Inc, Pembroke Pines, Florida
  - Mount Sinai, New York, New York
  - Penn State University Milton S. Hershey Medical Center, State College, Pennsylvania
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Envision Clinical Research, LLC, Laredo, Texas
  - Sagact, Pllc, San Antonio, Texas
- Bulgaria (6):
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - MHAT - Pazardzhik AD, Pazardzhik
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - MHAT "Sv. Karidad", EAD, Plovdiv
  - MHAT - Silistra AD, Silistra
  - MHAT "Sv. Petka" - Vidin, AD, Vidin
- Canada (2):
  - Brandon Medical Arts Clinic, Brandon, Manitoba
  - Humber River Hospital, Toronto, Ontario
- France (6):
  - CHU Amiens - Hopital Sud, Service d'Hépato-Gastroentérologie, Amiens
  - Cabinet Médical de Gastro-entérologie Dr.Lesage, Armentières
  - Hôpital Claude Huriez - CHU Lille, Service des maladies de l'appareil digestif, Lille
  - Cabinet Médical de Gastroentérologie Dr. Bismuth, Lille
  - Cabinet Médical de Gastroentérologie Dr. Ben Ali, Roubaix
  - Cabinet Médical de Gastro-entérologie Dr.Vernier Massouille, Tourcoing
- Hungary (7):
  - Principal SMO Kft., Baja
  - Semmelweis Egyetem, Budapest
  - Endomedix Diagnosztikai Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bugat Pal Korhaz, Gasztroenterologia, Gyöngyös
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Gastroenterologiai Osztaly, Kaposvár
  - Mazso-Pharma Kutatasfejlesztesi Kft, Szeged
- Italy (4):
  - Fondazione IRCCS Ospedale Maggiore, Policlinico Mangiagalli e Regina Elena. Dipartimento di Medicina e Specialità Mediche, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Dipartimento di Medicina Interna, Roma
  - Policlinico Universitario Agostino Gemelli, UOC Medicina Interna e gastroenterologia - CIC, Rome
- Latvia (5):
  - Polana D LLC, Daugavpils
  - J.Seleznovs Doctor Practice, Jelgava
  - Health Center 4, Affiliate Diagnostic Center, Riga
  - Riga East Clinical University Hospital, Riga
  - Pauls Stradins Clinical University Hospital SLLC, Riga
- Poland (5):
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Korczowski Bartosz, Gabinet Lekarski, Private Pediatric Office, Rzeszów
  - Niepubliczny Zaklad Opieki Zdrowotnej SONOMED, Szczecin
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - Ars-Medica S.C Rybak Maria, Rybak Zbigniew, Wroclaw
- Slovakia (3):
  - Alian s.r.o., Bardejov
  - B+B MED, s.r.o., Gastroenterologicka ambulancia, MUDr. Brandeburova, Košice
  - Gastromedic, s.r.o, Nové Zámky
- Ukraine (11):
  - Med Center of Eurolab LLC Policlinic Outpatient Dept O.O.Bogomolets NMU, Kyiv
  - CI of Kyiv RC Kyiv Regional Clinical Hospital, Kyiv
  - Lviv Regional Clinical Hospital D.Halytskyi Lviv NMU, Lviv
  - Lviv Municipal City Clinical Hospital #5 Dept of Therapy D.Halytsky Lviv NMU, Lviv
  - CI Odesa Regional Clinical Hospital, Center of Gastroenterology, Odesa
  - CI of SRC Sumy RCH Dept of Gasroenterology Sumy SU MI,Chair of Internal Medicine of PGE, Sumy
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Vinnytsya RCH for Patriotic War Invalides Therapeutic Dept # 1 Vinnytsia M.I.Pyrogov NMU, Vinnytsia
  - CI City Clinical Hospital #6 Dept of Gastroenterology, Zaporizhzhia
  - CI City Hospital #1, Dept of Surgery, Zaporizhzhia
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient IN: 28 November 2016 ; Last patient OUT: 31 July 2017
Pre-assignment Details: The study consisted of 3 phases:
  * Screening Phase - up to 4 weeks
  * Double-blind Placebo-controlled Phase - Weeks 0 to 8
  * Follow-up Phase - Week 9
Period: Overall Study
Arm/Group | 80 mg BID | 160 mg BID | Placebo
Started | 4 | 8 | 7
Completed | 2 | 2 | 4
Not Completed | 2 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 mg BID | 160 mg BID | Placebo | Total
Number analyzed (Participants) | 4 | 8 | 7 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 7 | 19
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 2 | 3 | 5 | 10
  Male | 2 | 5 | 2 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 7 | 6 | 17
  Black or African American | 0 | 1 | 0 | 1
  Not reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy on Ulcerative Colitis Disease Activity Index
Description: After 17 months, only 19 patients out of the target 207 patients, were enrolled in the study. Therefore neither descriptive nor comparative analyses were performed on outcome measures and the project in mild to moderate ulcerative colitis has been terminated.
Time Frame: up to 8 Weeks
Population: After 17 months, only 19 patients out of the target 207 patients, were enrolled in the study. Therefore neither descriptive nor comparative analyses were performed on outcome measures and the project in mild to moderate ulcerative colitis has been terminated
Groups:
- 80 mg BID: 80 mg BID treatment group
- 160 mg BID: 160 mg BID treatment group
- Placebo: Placebo treatment group
Arm/Group | 80 mg BID | 160 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- 80 mg BID: GED-0507-34-Levo 80 mg BID
- 160 mg BID: GED-0507-34-Levo 160 mg BID
- Placebo: Placebo treatment
Arm/Group | 80 mg BID | 160 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 1/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg BID (N=4) | 160 mg BID (N=8) | Placebo (N=7)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — worsening of ulcerative colitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT02808390/Prot_SAP_000.pdf